CLINICAL TRIAL: NCT02568228
Title: Health Beneficial Effects of Krill Oil and Lean and Fatty Fish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Olympic Seafood AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2015/706/REK sør-øst C
Record Dates: First submitted 2015-08-31; First posted 2015-10-05 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Triacylglycerols; Omega-3 fatty acids; Krill oil; Fish; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Krill group (Experimental): Krill oil capsules. 4 g/day encapsulated krill oil (Rimfrost Sublime) corresponding to ~900 mg/day EPA + DHA + DPA for 8 weeks. The participants will be instructed to take the capsules with the breakfast and dinner meals.
  Interventions: Dietary Supplement: Krill oil
- Fish group (Experimental): Lean and fatty fish. Three weekly test-meals, containing two meals of fatty fish and one meal of lean fish for 8 weeks corresponding to ~900 mg/day EPA + DHA + DPA.
  Interventions: Other: Lean and fatty fish
- Control group (Placebo Comparator): Placebo capsules. 4 g/day encapsulated high oleic sunflower oil (HOSO) for 8 weeks. The participants will be instructed to take the capsules with the breakfast and dinner meals.
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Krill oil — The krill group and the control group will be double blinded. The krill oil and placebo capsules will be administered in equal amounts and are of equal size and have the same color.
  Other Names: Rimfrost Sublime
  Arms: Krill group
Other: Lean and fatty fish — The fish group will be open labeled.
  Arms: Fish group
Dietary Supplement: Placebo capsules — The krill group and the control group will be double blinded. The krill oil and placebo capsules will be administered in equal amounts and are of equal size and have the same color.
  Arms: Control group

SUMMARY:
Intake of omega-3 (n-3) polyunsaturated fatty acids (PUFAs) from fish oil and fish are associated with significant health benefits in risk of cardiovascular disease. However, both lean and fatty fish have been shown to have beneficial effects suggesting that not all effects are mediated by n-3 PUFAs. Krill oil is an n-3 PUFA supplement on the marked. The n-3 PUFAs from krill oil is in the form of phospholipids, and these fatty acids may be more readily and effectively absorbed after ingestion than n-3 PUFAs in the form of triacylglycerols from fish oil. Fish also contain many other potential health components than n-3 PUFAs such as taurine and vitamin D, iodine, selenium and more unspecified components such as bioactive peptides which can mediate the health beneficial effects observed after intake of fish.

The present study aims to elucidate the cardiovascular health beneficial effects after consumption of fish (lean and fatty) and krill oil, with regard to effects on plasma lipids and other markers of cardiovascular health such as inflammatory, haemostatic and endothelial dysfunction markers. The investigators will perform whole genome transcriptome analyses in peripheral blood mononuclear cells (PBMCs) in order to further understand the cardiovascular health benefits and elucidate the mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (CRP < 10 mg/L)
* Stable weight (± 5 % of body weight) the last three months
* BMI 18.5-35 kg/m2
* Fasting triglycerides 1.3-4.0 mmol/L
* Willingness to eat fish
* Willingness to not take omega-3 or other dietary supplements during the study.

Exclusion Criteria:

* Pregnancy or lactation
* Any chronic disease, including diabetes type 1 or 2. CVD or cancer past 6 months
* Elevated thyroid hormones or TSH levels
* Elevated total cholesterol (>7.8 mmol/L) or fasting triglycerides (>4.0 mmol/L)
* Use of prescription drugs that may affect triglycerides (e.g. diabetes drugs, Cyclosporin A, Orlistat and Sibutramine), except statins if stable dose past 3 months.
* Blood pressure > 160/100 mmHg
* Hormone treatment (except stable doses the past three months of contraceptives or thyroxine)
* Planned weight loss
* The use of Vita Proactive or other food items enriched with plant sterols
* Excessive alcohol consumption (>40 g/day)
* Habitual fish consumption of more than one serving of fatty fish per week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Fasting triglycerides | 8 weeks

SECONDARY OUTCOMES:
Circulating inflammatory markers | 8 weeks
  Such as TNFalpha and IL-6
Gene expression of inflammatory markers and genes in lipid metabolism | 8 weeks
  Measured with RT-qPCR
Plasmamlipids | 8 weeks
  Such as total- LDL- and HDL-cholesterol
Lipoprotein subclasses | 8 weeks
Plasma fatty acid composition | 8 weeks
Blood pressure | 8 weeks
Endothelial dysfunction markers | 8 weeks
  Sush as NOx and ADMA
Hemostatic markers | 8 weeks
  Such as vWF and thrombomudulin
Muscle strength | 8 weeks
  Measured by hand grip strength and chair stand test
Whole genome transcriptome analysis in PBMC | 8 weeks
  Changes in the gene expression profile
Metabolome profile in blood | 8 weeks
  In blood
Metabolome profile in urine | 8 weeks
  In urine

CONTACTS AND LOCATIONS:
Overall Officials: Stine M Ulven, PhD, Principal Investigator — University of Oslo